CLINICAL TRIAL: NCT00187837
Title: The CAP-1 Trial: Effect of Stepwise Versus One Completed Excavation in Deep Caries in Permanent Teeth: A Randomised, Patient - and Observer-blinded Multicenter Trial
Brief Title: The CAP-1 Trial: Stepwise Excavation Versus One Completed Excavation in Deep Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: National Health Insurance foundation (Unknown); Dan Dental A/S (Industry); University of Aarhus (Other); Göteborg University (Other); Huddinge Faculty,Stockholm,Sweden (Unknown); Uppsala FolkTandvård,Sweden (Other); Malmö Dental school,Sweden (Unknown)
Responsible Party: Principal Investigator, Lars Bjørndal, PhD, Dr. Odont, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10001
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Dental Caries; Reversible Pulpitis
Keywords: Stepwise excavation
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SW intervention (Experimental): Stepwise Excavation
  Interventions: Procedure: SW
- DCE intervention (Other): Control intervention Direct complete excavation. The updated terminology for completed excavation is non-selective excavation to hard dentin
  Interventions: Procedure: DCE

INTERVENTIONS:
Procedure: SW — Stepwise removal of carious tissue in 2 stages
  Other Names: Stepwise carious removal wos
  Arms: SW intervention
Procedure: DCE — one complete excavation
  Other Names: Non-selective carious removal to hard dentin
  Arms: DCE intervention

SUMMARY:
Brief summary

Background:

A large proportion of dental practice involves the treatment of caries in the permanent dentition. In USA alone tooth related pain is annually responsible for 15 billions days lost through sickness. We do not know whether a stepwise excavation is better or worse compared with one final completed excavation in adults with deep caries with or without pain. A deep carious lesion is in the risk zone of being pulpal exposed during excavation.

Aim:

The aim of the CAP-1-trial is to investigate the beneficial effects of stepwise excavation during two visits versus óne completed excavation of deep caries in permanent teeth with or without pain.

Patients:

Consecutive patients contacting the units involved in the CAP trial for the treatment of deep caries. The trial will comprise 300 patients.

Design:

CAP-1-trial is a randomised patient- and observer-blinded multicenter trial, with two parallel intervention groups. Patients that fulfill the inclusions criteria and none of the exclusions criteria, will be centrally bloc-randomised in Copenhagen Trial Unit, Copenhagen DK, and stratified by age and pain. Allocation ratio is 1:1.

Interventions and products:

Patients are allocated for stepwise excavation in two visits or final excavation in one visit. The patients will not be informed about the result of the randomisation, i.e. the type of intervention. Therefore, all patients will be contacted for two visits. The second visit in the stepwise excavation group wil be used for the second and final excavation, and for the performance of a permanent restoration. The second visit in the one step excavation group will solely be used for the performance of a permanent restoration. The interventions in both groups are completed following 8-10 weeks after the randomisation.

A temporary calcium hydroxide based material is used in both groups (Dycal®). The temporary restoration material, glas-ionomer cement is used (Ketac Molar®) in between visits, and a resin material is used for the final restoration(Herculite®).

DETAILED DESCRIPTION:
References

BJERKÉN E, WENNBERG A, TRONSTAD L. Endodontisk akutbehandling. Tandläkartidningen. 1980;72:314-9.

BJØRNDAL L, REIT C. The annual frequency of root-fillings, tooth extractions and pulp related procedures in Danish adults 1977-2003. Int Endod J 2004:37:782-788.

BJØRNDAL L. The deep caries lesion dilemma. In Nordic Dentistry 2004 yearbook (Schou L, ed). Copenhagen, Denmark: Quintessence Publishing Co, Inc., 2004; 107-20.

BJØRNDAL L & THYLSTRUP A. A practice -based study on stepwise excavation of deep carious lesions in permanent teeth: a 1-year follow-up study. Community Dent Oral Epidemiol 1998;26:122-8.

BJØRNDAL L. Treatment of deep carious lesions with stepwise excavation. A practice-based study. Tandlaegebladet 1999;103:498-506.

BJØRNDAL L, LARSEN T, THYLSTRUP A. A clinical and microbiological study of deep carious lesions during stepwise excavation using long treatment intervals. Caries Res 1997;31:411-.

BJØRNDAL L, LARSEN T. Changes in the cultivable flora in deep carious lesions following a stepwise excavation procedure. Caries Res 2000;34:502-8.

BERGENHOLTZ G, SPÅNGBERG L. Controversies in endodontics. Crit Rev Oral Biol Med 2004;15:99-114.

FOUAD AF. Molecular mediators of pulpal inflammation. In Seltzer and Bender's Dental pulp ( Hargreaves KM, Goodis HE, eds). Chicago, USA: Quintessence Publishing Co, Inc., 2002; 247-79.

KARLSSON P-O, REIT C. Reasons for endodontic treatment among Swedish general practitioners (abstract). Int Endod J 1994;27:100.

KIRKEVANG L-L Periapical and endodontic status in Danish populations (Ph.D: thesis). Århus: University of Aarhus; 2001.

LEKSELL E, RIDELL K, CVEK M, MEJÁRE I. Pulp exposure after stepwise versus direct complete excavation of deep carious lesions in young posterior permanent teeth. Endod Dent Traumatol 1996;12:192-96.

MAGNUSSON B, SUNDELL SO. Stepwise excavation of deep carious lesions in primary molars. J Int Ass Child 1977;8:36-40.

NADIN G, GOEL BR, YEUNG Ca, GLENNY AM. Pulp treatment for extensive decay in primary teeth (Cochrane Review). In: The Cochrane Library, Issue 1, 2004. Chichester,Uk: John Wiley & Sons, Ltd.

NÄRHI M. Dentinal and pulpal pain. In Textbook of Endodontology (Bergenholtz G, Hørsted-Bindslev P, Reit C, eds). Oxford, UK: Blackwell Munksgaard, 2003; 43-56.

REIT C, HEDEN G, MILTHON R. Endodontiskt behandlingspanorama inom allmäntandvården. Tandläkartidningen 1993;85:543-6.

RICKETTS DNJ, KIDD EAM, INNES N. Complete or ultraconservative removal of decayed tissue in unfilled teeth (Protocol for a Cochrane Review). In: The Cochrane Libray, Issue 1, 2004. Chichester , UK: John Wiley & Sons, Ltd.

SJÖSTRÖM O, SUNDBERG H. Arbetstidens fördelning på olika verksamheter i svensk tandvård 1988. Tandläkartidningen 1989;81:856-67.

SUDA H, IKEDA H. The circulation of the pulp. In Seltzer and Bender's Dental pulp (Hargreaves KM, Goodis HE, eds). Chicago, USA: Quintessence Publishing Co, Inc., 2002; 123-50.

TAYLOR H, CURRAN NM. The Nuprin Pain Report. New York, Lou Harris, 1985.

ELIGIBILITY:
Inclusion Criteria:

* Person ≥ 18 yrs having deep caries with or without pain:
* x-ray show primary caries in the inner 1/4 of the dentin, with the presence of a radiopaque zone at the pulpal wall NB: Need to mark a 'yes' for both criteria!

Exclusion Criteria:

* Deep carious tooth with (irreversible pulpitis)unbearable pain and/or disturbed night's sleep)
* Deep carious tooth negatively responding on thermal and electrometric tests.
* Deep carious tooth has 'attachment loss' > 5 mm
* X-ray shows apical radiolucency of the actual tooth
* Deep carious tooth has restoration in direct contact with the pulp
* The person has problems with communication
* No informed and written consent is present
* Due to health conditions or pregnancy the person can not participate in the trial

NB: Need to mark 'No' for all criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2005-02; Primary Completion 2007-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome is whether the treatment can be made with a maintained sensible pulp and without root infection following a 1-year control. | 1year control data for all treatments primo 2008
  In this update we have also completed 5 yr control

SECONDARY OUTCOMES:
Secondary outcome constitutes pain intensity using a visual analogue scale measured before the first visit and 1 and 7 days after. | ultimo 2007

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bjørndal, Study Director — University of Copenhagen
Locations (1):
- School of Dentistry, Faculty of Health Sciences, Copenhagen, Copenhagen N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
1½ yr results published in European Journal of Oral Sciences 2010; 118: 290-297.

REFERENCES:
- [Result] Bjorndal L, Reit C, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Thordrup M, Dige I, Nyvad B, Fransson H, Lager A, Ericson D, Petersson K, Olsson J, Santimano EM, Wennstrom A, Winkel P, Gluud C. Treatment of deep caries lesions in adults: randomized clinical trials comparing stepwise vs. direct complete excavation, and direct pulp capping vs. partial pulpotomy. Eur J Oral Sci. 2010 Jun;118(3):290-7. doi: 10.1111/j.1600-0722.2010.00731.x. PMID 20572864
- [Derived] Bjorndal L, Fransson H, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Hedenbjork-Lager A, Dige I, Thordrup M. Randomized Clinical Trials on Deep Carious Lesions: 5-Year Follow-up. J Dent Res. 2017 Jul;96(7):747-753. doi: 10.1177/0022034517702620. Epub 2017 Apr 14. PMID 28410008